CLINICAL TRIAL: NCT05699889
Title: Prevalence of COVID-19-associated Kidney Injury in ICU and Prognosis of Proximal Tubular Injury in ARDS: the URICOV Study
Brief Title: Acute Kidney Dysfunction in COVID-19 and Non-COVID-19 Related ARDS
Acronym: URICOV
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM20_0177
Record Dates: First submitted 2023-01-24; First posted 2023-01-26 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Acute Kidney Injury Due to COVID-19
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients in intensive care for SARS-CoV 2 infection with severe respiratory impairment.
  Interventions: Other: Data collection
- Patients in intensive care without SARS-CoV 2 infection with severe respiratory impairment.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — acute kidney injury and tubular dysfunction

SUMMARY:
In addition to respiratory involvement, SARS-CoV 2, the virus responsible for coronavirus 2019 or Covid-19, appears to be responsible for renal involvement such as acute renal failure or proteinuria, so the mechanisms are not known at this time. The consequences of Covid-19 on renal function in the short and long term are not known.

It is important to be able to better document these renal impairments to understand the mechanisms of this disease.

The main objective of this study is to describe the prevalence of Covid-19-related renal damage (acute renal failure, proteinuria, microalbuminuria, hematuria) in a large cohort of patients in intensive care for SARS-CoV 2 infection with severe respiratory impairment.

The other objectives will be to evaluate in this cohort the impact of these renal impairments on the severity of the Covid-19 disease, and to compare them to the renal impairments of patients in intensive care for acute respiratory distress syndrome (ARDS) due to other respiratory diseases.

Blood and urine samples will be taken at the time of intubation in all critically ill patients with respiratory distress requiring mechanical ventilation for Covid-19 or other cause of respiratory distress with PaO2/FiO2 ratio < 300.

Patients will be followed for the duration of their ICU and hospital stay. Data will be collected prospectively in three ICUs in the University Hospitals of Marseille.

ELIGIBILITY:
Inclusion Criteria:

* • Displaying acute respiratory distress Needing invasive mechanical ventilation

  * With PaO2/FiO2 ratio < 300 after orotracheal intubation

Exclusion Criteria:

* Patients in ICU following thoracic surgery or lung transplantation
* Patients with cardiogenic pulmonary oedema
* Patients with end stage kidney disease
* Moribund patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in intensive care for SARS-CoV 2 infection with severe respiratory impairment and Patients in intensive care without SARS-CoV 2 infection with severe respiratory impairment
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the incidence of acute kidney injury and tubular dysfunction | First 24 hours after orotracheal intubation
  We aimed to perform a detailed analysis of urinary markers of kidney dysfunction with urine protein electrophoresis and tubular protein dosage in a prospective cohort of critically ill patients in ICU for ARDS due to COVID-19 in the first 24 hours following orotracheal intubation, to evaluate the incidence of acute kidney injury (AKI) and tubular dysfunction among critically ill patients with COVID-19-related ARDS at the onset of Mechanical ventilation, and to specify which part of the kidney parenchyma is involved.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie GARRIDO-PRADALIE, Study Director — Assistance Publique Hopitaux De Marseille; Mickaël BOBOT, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France